CLINICAL TRIAL: NCT04538534
Title: Nicardipine to Avoid Spasm in Trans Radial Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pr. Semir Nouira (Other)
Responsible Party: Sponsor-Investigator, Pr. Semir Nouira, MD, University of Monastir
Organization: University of Monastir (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TN2020-NA T -INS-39
Record Dates: First submitted 2020-05-31; First posted 2020-09-04 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Spasm Artery
Keywords: radial artery spasm
MeSH Terms: interventions — Nicardipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nicardipine and isosorbide dinitrate (Experimental): A Cocktail of 1 mg of Isosorbide Dinitrate associated to 1 mg of nicardipine will be put in a syringe than diluted in saline serum to have a volume of 3cc.
  The obtained solution will be administered in an intra-arterial fashion via the trans-radial sheath after randomization.
  Interventions: Drug: Nicardipine
- isosorbide dinitrate (Active Comparator): Isosorbide Dinitrate: 1 mg will be diluted in saline solution as to have a 3cc volume The obtained solution will be administered in an intra-arterial fashion via the trans-radial sheath after randomization
  Interventions: Drug: Nicardipine

INTERVENTIONS:
Drug: Nicardipine — To compare the association of nicardipine and isosorbide dinitrate vs isosorbide dinitrate alone on the rate of occurrence of radial artery spasm
  Other Names: Loxen

SUMMARY:
Radial artery is the recommended route for percutaneous coronary intervention for it significantly reduces net adverse clinical events compared to the femoral approach. The success of the radial approach is therefore of a paramount importance. However, radial artery spasm (RAS) remains one of the major limitations of transradial approach (TRA) and the most frequent cause of TRA failure. Several recommendations has been issued to improve success rate when using the radial route.

In the Tunisian difficult economic context, the use of low end equipment, the unavailability of nitroglycerine and calcium antagonist verapamil, has led to the general feeling that RAS and TRA failure has subsequently increased.

The standard and only used protocol by the Tunisian interventional cardiologist, consists of administrating 1 mg isosorbide dinitrate through the arterial sheath immediately after radial arterial puncture, therefore limiting the options to prevent RAS.

Nicardipine is the only injectable calcium antagonist available in Tunisia. Its spasmolytic action on radial artery has been well demonstrated when used in CABG. However, it has been very poorly investigated in trans radial percutaneous coronary intervention.

Investigators believe that the concomitant use of nicardipine with isorbide might significantly reduce RAS and TRA failure when compared to isosorbide dinitrate only.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for coronary intervention will be eligible for screening (coronarography or coronary angioplasty).
* Participant is willing and is able to give informed consent for participating in the trial.
* Male or Female, aged 18 years or above.

Exclusion Criteria:

* Planned femoral approach because no radial pulse was perceived
* Cardiogenic shock
* Coronary intervention for ST elevation myocardial infarction during the night shift.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants in which radial artery spasm occurred | 24 hours
  Significant limitation of the catheter movement perceived by the operator together with mild to severe pain in the forearm of the patient or the need of repeating vasodilator administration

SECONDARY OUTCOMES:
Number of Participants in which severe radial artery spasm occurred | 24 hours
  Complete catheter blockage [i.e., the catheter cannot be moved back or forth], severe pain with need for morphine or midazolam injections, crossover to the contralateral radial or femoral artery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Fattouma Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No